CLINICAL TRIAL: NCT05610527
Title: Targeting the Knowledge Gap for Sex-specific Hormonal Influences on Inflammatory Bowel Disease Symptoms and Management
Brief Title: Hormonal Influences on Inflammatory Bowel Diseases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: IRB_00160085
Record Dates: First submitted 2022-10-13; First posted 2022-11-09 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Inflammatory Bowel Diseases; Contraception; Menstrual Problem
Keywords: randomization; inflammatory markers; patient reported outcome measures
MeSH Terms: conditions — Inflammatory Bowel Diseases; Menstruation Disturbances | interventions — Restraint, Physical

STUDY DESIGN:
Intervention Model Description: Prospective cohort study of females with IBD: 100 hormonal contraceptive users and 100 naturally cycling participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hormonal contraception users (Active Comparator): Females with inflammatory bowel disease who use hormonal contraception (combination oral contraceptives, the etonogestrel implant, or the levonorgestrel intrauterine device)
  Interventions: Other: Proposed study design and randomization scenarios; Other: Repeated measures of validated Inflammatory Bowel Disease Patient Reported Outcome Instruments; Other: Inflammatory marker collection and assessment for correlation with PRO responses and menstrual timing
- Naturally cycling participants (Other): Females with inflammatory bowel disease who do not use hormonal contraception and have regular menstrual cycles (self or partner permanent contraception, copper IUD, abstinence, barrier methods, and fertility awareness methods)
  Interventions: Other: Proposed study design and randomization scenarios; Other: Repeated measures of validated Inflammatory Bowel Disease Patient Reported Outcome Instruments; Other: Inflammatory marker collection and assessment for correlation with PRO responses and menstrual timing

INTERVENTIONS:
Other: Proposed study design and randomization scenarios — Present hypothetical study scenarios and assess willingness to be randomized based on the adapted 7-item Attitudes to Randomized Trials Questionnaire
Other: Repeated measures of validated Inflammatory Bowel Disease Patient Reported Outcome Instruments — We will electronically administer Ulcerative Colitis (UC) and Crohn's Disease validated PRO instruments, including the daily symptom modules and weekly quality of life modules for 12 weeks to all 200 participants
  Other Names: UC PRO Instrument; Crohn's PRO Instrument
Other: Inflammatory marker collection and assessment for correlation with PRO responses and menstrual timing — In an Aim 3 sub study of 30% of participants, we will collect inflammatory markers commonly used to assess disease activity and risk of relapse in inflammatory bowel disease patients, including weekly blood samples of high sensitivity c-reactive protein (13 total) and monthly ferritin, albumin, and WBC, as well monthly stool specimens (4 total) for fecal calprotectin
  Other Names: Inflammatory markers

SUMMARY:
Of the 1.8 million females with inflammatory bowel diseases (IBD) in the US, over half of those who are premenopausal suffer from cyclical menstrual-related IBD symptoms, regardless of how well their disease is controlled. Despite the significant impact that cyclical IBD symptoms, such as abdominal pain, diarrhea, and fatigue have on quality of life, evidence about how to alleviate these symptoms is lacking. In other chronic conditions which are hormonally influenced, such as epilepsy, hormonal contraception may be used to favorably impact disease-related symptoms associated with menses and improve quality of life. In our previous cross-sectional study, 47% of the levonorgestrel intrauterine device users and 19% of combination oral contraceptive users reported improvement in their cyclical IBD symptom. All hormonal methods may plausibly improve symptoms, but prospective, rigorous data evaluating their efficacy for this purpose are lacking. In order to design a future comparative effectiveness trial on the effect of hormonal contraceptive methods on menstrual-related IBD symptoms, we propose this pilot prospective cohort study of 200 females with IBD: 100 naturally cycling and 100 hormonal contraception users. We will gain essential knowledge on IBD-specific influences on contraceptive method selection, willingness to be randomized to methods, the ability of IBD patient reported outcome (PRO) instruments to differentiate between non-menstrual and menstrual-related IBD symptoms, and assess the potential role of inflammatory markers as outcome measures in future trials. We will recruit participants from the University of Utah IBD Center and clinics, other Utah gastroenterology providers, and through social media ads. Total study commitment will be ~12 weeks. Study activities will include daily and weekly text message surveys, as well as blood draws and fecal samples for inflammatory markers in a subset of participants which are commonly used for IBD management. Our aims include: (1) To identify preferences and reasons for contraceptive method selection (or non-use) and willingness to participate in a randomized controlled trial, to inform feasibility of a future trial, (2) To obtain estimates of means and standard deviations for the validated Crohn's Disease and Ulcerative Colitis PRO Instruments by menstrual timing in naturally-cycling participants and between bleeding and non-bleeding days in hormonal contraception users, and (3) To assess correlation between inflammatory marker changes (fecal calprotectin & high sensitivity C-reactive protein), menstrual timing or bleeding/non-bleeding days, and IBD PRO responses, in a subset of 30% of Aim 1 participants. This pilot will inform a future trial design to define non-contraceptive benefits of hormonal contraception on cyclical IBD symptoms. This line of inquiry will allow for an adjuvant approach for IBD symptom management that is sex-specific and addresses both concerns for hormonal triggers and the need for highly-effective contraception for those who desire it.

DETAILED DESCRIPTION:
Aim 1. Identify preferences and reasons for contraceptive method selection (or non-use) and willingness to participate in a future randomized controlled trial in 200 participants with IBD (100 naturally cycling and 100 hormonal contraception users). Our a priori cut off requires ≥ 75% of participants accepting randomization.

Hypothesis: The majority of participants will accept randomization if they may switch methods if not satisfied.

Aim 2. Obtain estimates of means and standard deviations for the validated Crohn's Disease and Ulcerative Colitis PRO Instruments across the menstrual cycle (menses, ovulation, pre-menstrual) in the naturally-cycling participants and between bleeding and non-bleeding days in the hormonal contraception users.

Hypothesis: IBD PRO instruments will reliably reflect IBD symptom changes related to menstrual phases.

Aim 3. Assess the correlation between inflammatory marker changes (fecal calprotectin & high sensitivity C-reactive protein), menstrual timing and/or bleeding days, and IBD PRO responses in a subset of 30% of Aim 1 participants (30 naturally cycling and 30 hormonal contraception users).

Hypothesis: Changes in inflammatory markers will be correlated with menstrual phases and IBD PRO responses.

Study Design: A pilot prospective cohort study of 200 women with IBD (100 naturally cycling and 100 hormonal contraception users).

Recruitment. We will recruit via four different sources: 1. With the support of the co-investigators who are IBD subspecialists at the University of Utah (Drs. Flynn and Johnson), we will send recruitment emails to their patients who meet inclusion criteria via the Epic patient portal (MyChart). 2. We will post fliers regarding the study in the gastroenterology, primary care, and women's health clinics across University of Utah sites. 3. We will send recruitment materials to other non-university gastroenterology sites in Utah. 4. We will advertise via social media nationally with a link to a University of Utah Research Enterprise Data Capture (REDCap) survey to assess eligibility and provide contact information for study coordinators to connect for a phone screen.

AIM 1 Sample Size: This is a pilot study designed to collect baseline data to inform future trials and not powered to assess statistical differences between study groups. We plan to recruit 200 participants in an IBD setting who represent common contraceptive method choices and compare hormonal method users to non-users regarding preferences in method selection. The sample size will also give a breadth of perspectives on willingness to be randomized to different hormonal methods under variable study conditions and designs to influence a future trial. Our sample size takes into consideration feasibility for recruitment given our recruitment timeline, as well as sample size recommendations for pilot clinical trials.

Participant procedures: Total study engagement is 12 weeks. Enrollment processes. Study staff will complete a phone screening, discuss study procedures, and if they meet inclusion criteria, either email the potential participant the consent and enrollment survey for completion via REDCap or schedule an in-person enrollment visit if participating in the Aim 3 sub study to allow for inflammatory marker collection. The screening phone call will include request of documentation confirming IBD diagnosis and screening questions regarding timing of IBD diagnosis, current disease activity, prior endoscopy and surgery dates, current and prior treatments, and any hospitalizations. These responses and documentation of diagnoses will be reviewed for eligibility by the IBD subspecialists before consent and enrollment is completed.

Survey content. The enrollment survey will assess sociodemographic and reproductive characteristics, IBD history as above, menstrual cycle timing and symptoms including bleeding characteristics and pain scores, sexual satisfaction surveys, baseline IBD symptom PRO instruments, menstrual-related IBD symptoms, prior and current contraceptive experiences, and preferences regarding contraceptive methods. Using an adapted 7-item Attitudes to Randomized Trials Questionnaire, participants will be presented with hypothetical RCT scenarios to assess willingness to be randomized based on different methods, different study designs (e.g. participant preference arm), options to switch methods, and then query regarding reasoning if not willing to be randomized.

Study Arms: The "naturally-cycling" cohort will include participants who are not using any form of hormonal contraception and meet inclusion criteria with regular menses. This may include non-hormonal method users, including abstinence, copper IUD, self or partner permanent contraception, barrier methods, or fertility awareness methods. The hormonal contraception user cohort includes the most common hormonal contraceptive options (COC, LNG IUD, ENG implant). The hormonal contraceptive method must have been initiated prior to study enrollment, thus the method choice made outside of this study is not an intervention. If a participant initiates, stops, or switches methods during the study, they will be analyzed in the assigned cohort at enrollment, as changes in hormonal methods may not result in consistent bleeding profiles or resumption of natural cycles for weeks to months.

Follow-up. While the aim 1 outcome assessment occurs with the enrollment survey, all participants will be followed for Aim 2 and a subset for Aim 3 for 12 weeks from the time of enrollment. Participants will receive compensation for time with each completed study activity.

Analyses. The goal of Aim 1 is to define the characteristics of the IBD study population and determine a point estimate of the proportion of participants willing to be randomized to one of three contraceptive methods under each scenario characteristics. A 95% confidence interval around this estimate will describe its variability. The 7-item Attitudes to Randomized Trials Questionnaire30 is not scored in sum, but each item adds characteristics related to the proposed study design that are reported via descriptive statistics as positive or negative attributes influencing randomization willingness. We will report contraceptive method preferences and IBD-specific reasons for method selection (and non-use of hormonal methods) via descriptive statistics, inferential analysis exploring relationships between respondent characteristics and method preferences, adjusting for participant characteristics as well as thematic findings from free text response options. For free text responses, we will use frequency distributions as well as Latent Dirichlet Allocation, a topic modeling technique to identify common themes and patterns in the responses. We will also conduct comparative analysis to compare IBD-specific reasons for method selection or non-use of hormonal methods across different demographics and disease characteristics. While the enrollment survey and all daily and weekly PRO instruments will be administered electronically to all participants, we anticipate that certain significant differences may also exist between participants who agree to enroll in Aim 3 and those who do not. This may be due to their willingness to come for in-person lab assessments and engagement with the study team. We will thus perform sensitivity analyses to determine, for each of these groups, the proportion willing to be randomized and to assess contraceptive method preferences. Similarly, we will perform sensitivity analyses for both those who switch, discontinue or initiate a contraceptive method and for those who are abstinent and may be using hormonal contraception for non-contraceptive purposes only compared to those who need contraception for pregnancy prevention.

AIM 2 Sample size. All study participants recruited in Aim 1 will be included in this aim. We anticipate a 5% attrition in survey completion over 12 weeks.

Procedures. Participants will receive electronic survey links to assess IBD-related and menstrual-related symptoms, QOL measures, sexual activity and health changes across menstrual cycles and bleeding and non-bleeding days in the hormonal contraception users over 12 weeks. Via REDCap, we will send automated reminders and deliver links for data completion through text messages to the participant's mobile phone or device. Participant responses automatically upload from the phone or device to REDCap.

Daily surveys. Daily surveys will begin the day of enrollment and continue for 12 weeks. The survey questions include either the CD or UC PRO instrument depending upon diagnosis. The daily IBD PRO instruments include modules on signs and symptoms, systemic symptoms, and coping strategies with a total of 17 questions (6 minutes) for the CD PRO and 20 questions (7 minutes) for the UC PRO. We will also query chronic pelvic pain severity, vaginal bleeding and amount, and if bleeding, menstrual-related pain and severity (4 follow-up questions if bleeding).

Weekly Surveys. The weekly surveys will begin on day of enrollment and continue every week for 12 weeks (13 total with the enrollment survey). These longer surveys will include the daily questions plus the IBD PRO modules on daily life impact with 9 questions (3 minutes) and emotional impact with 8 questions (3 minutes). Participants will complete a Likert scale on how bothersome IBD symptoms have been in the past week, and report any sexual activity with assessment of dyspareunia, additional treatments for IBD or menstrual symptoms, and any changes to health history.

Analyses. This aim will assess changes in IBD PRO responses over subsequent menstrual cycles and between bleeding and non-bleeding days for hormonal contraceptive users. The UC PRO and CD PRO instrument modules will all be scored based on guidelines for instrument use. Report of bothersome IBD symptoms, chronic pelvic pain, dysmenorrhea, and dyspareunia will be on a Likert scale from 0-10. Any other reported changes in health, treatments or concerns will be reported by frequency and cycle timing. We will compare variations in these means across menstrual cycle timing using linear regression and compare means in symptom scores between cohorts using paired t-tests.

AIM 3 Sample size. We will enroll 30% of each cohort from Aim 1 in this sub study for a total of 60 participants.

Procedures. Potential participants eligible for Aim 1 who are willing and able to come to a study enrollment visit and 12 subsequent lab visits at the University of Utah will be offered participation in this Aim 3 sub study. For those interested, their enrollment will occur in-person, rather than virtually in order to initiate the inflammatory marker collection. At the enrollment visit, the research staff review the same electronic consents used for participants in Aim 1 and 2 and prompt completion of the enrollment survey using the University of Utah's secure, web-based REDCap system. The enrollment visit will also include urine pregnancy testing, lab testing (complete blood count, hsCRP, ferritin, and albumin) and they will receive a kit to collect fecal calprotectin from a home stool sample and return it at the 1-week blood draw. Lab assessments of inflammatory markers will occur at varying intervals. WBC, ferritin and albumin will be assessed at baseline screening visit and again monthly (4 total). The hsCRP will be measured at baseline and then occur weekly (13 total). Fecal calprotectin (from 1st morning stool) will be measured at baseline (sample collected at 1-week blood draw after enrollment) then monthly for 12 weeks (4 total). The blood draws and fecal calprotectin assessments that occur after the single in-person enrollment visit can be completed at local University labs throughout the region.

Analyses. We will compare the proportion of participants with hsCRP and fecal calprotectin levels within a 'normal' range by cohort (naturally cycling vs hormonal contraception users) using chi square. We will compare variations in means across menstrual cycles using mixed effects models. We will look for difference in inflammatory marker levels across IBD PRO responses and specific modules by including these PROs as covariates in our regression models, and will include a random intercept in our models for participants in order to account for variations in individual baseline marker levels.

ELIGIBILITY:
INCLUSION CRITERIA:

* Between 18-45 years old
* Fluent in English and/or Spanish
* Have biopsy-proven UC or CD (confirmed by medical records and/or through screening questions- see below enrollment procedures Aim 1)
* Willing to comply with study activities
* Have a reliable smartphone or text-message capable device for e-diary reminders and completion
* Regular menses (21-35d) when not on hormonal contraception
* For the hormonal contraception cohort, use of the LNG IUD, ENG implant, or COC
* For the naturally-cycling cohort, use of any non-hormonal method of contraception, including: self or partner permanent contraception, copper IUD, abstinence, barrier methods, and fertility awareness methods

EXCLUSION CRITERIA:

* Current pregnancy
* Breastfeeding without resumption of 2 normal menses
* Desires starting, stopping or switching hormonal contraception during the 12-week study timeframe
* History of hysterectomy
* Menopausal (no menses for 12+months when not on hormonal contraception
* Use of systemic gender-affirming hormone therapy (e.g. testosterone)
* Indeterminant or microscopic colitis
* Participation in any other clinical trials during this study timeline

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Must have menstrual cycles
Enrollment: 200 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Willingness to be randomized and reason and preferences for contraceptive method selection in the setting of IBD | Collected on enrollment survey
  Proportion of participants willing to be randomized in each hypothetical study scenario based on the adapted 7-item Attitudes to Randomized Trials Questionnaire and Proportion of participants who select each hormonal methods vs non-hormonal and characteristics as desirable
Change in IBD PRO responses/scores and by menstrual timing in natural cycling and bleeding vs non-bleeding days in hormonal contraception users | Daily symptom modules and weekly quality of life modules for 12 weeks
  UC PRO or CD PRO instrument scores by module. Modules 1-3 assess daily symptoms and modules 4-5 assess weekly quality of life measures.
Correlation in inflammatory marker changes to IBD PRO responses | Weekly blood draws (13 total) and monthly stool sample collection (4 samples)
  hsCRP and fecal calprotectin levels measured at baseline and at each collection visit throughout study UC PRO or CD PRO instrument scores by module. Measured daily or weekly on follow-up surveys.

SECONDARY OUTCOMES:
Acceptability and adherence to electronic PRO surveys | 12 weeks
  Proportion of participants who complete the daily and weekly survey assessments and rate acceptability of good to excellent on a 5-point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Lori Gawron, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No